CLINICAL TRIAL: NCT05594602
Title: A NON-RANDOMIZED, OPEN-LABEL, THREE-PART, DRUG-DRUG INTERACTION STUDY TO EVALUATE THE EFFECTS OF ITRACONAZOLE, CARBAMAZEPINE, AND QUINIDINE ON THE PHARMACOKINETICS AND SAFETY OF EDP-235 IN HEALTHY PARTICIPANTS
Brief Title: Drug-Drug Interaction Study Between EDP-235, Itraconazole, Carbamazepine and Quinidine in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EDP 235-002
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: drug-drug interaction
MeSH Terms: conditions — COVID-19 | interventions — EDP-235; Itraconazole; Carbamazepine; Quinidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-235 and Itraconazole interaction (Part 1) (Experimental): Subjects will receive EDP-235 and Itraconazole on respective dosing days
  Interventions: Drug: EDP-235; Drug: Itraconazole
- EDP-235 and Carbamazepine interaction (Part 2) (Experimental): Subjects will receive EDP-235 and Carbamazepine on respective dosing days
  Interventions: Drug: EDP-235; Drug: Carbamazepine
- EDP and Quinidine interaction (Part 3) (Experimental): Subjects will receive EDP-235 and Quinidine on respective dosing days
  Interventions: Drug: EDP-235; Drug: Quinidine

INTERVENTIONS:
Drug: EDP-235 — Subjects will receive EDP-235 on Days 1 and 14
  Arms: EDP-235 and Itraconazole interaction (Part 1)
Drug: EDP-235 — Subjects will receive EDP-235 on Days 1 and 23
  Arms: EDP-235 and Carbamazepine interaction (Part 2)
Drug: EDP-235 — Subjects will receive EDP-235 on Days 1 and 8
  Arms: EDP and Quinidine interaction (Part 3)
Drug: Itraconazole — Subjects will receive itraconazole QD Days 5-18
  Arms: EDP-235 and Itraconazole interaction (Part 1)
Drug: Carbamazepine — Subjects will receive carbamazepine BID Days 5-23 and Days 24-27
  Arms: EDP-235 and Carbamazepine interaction (Part 2)
Drug: Quinidine — Subjects will receive quinidine BID Days 5-12
  Arms: EDP and Quinidine interaction (Part 3)

SUMMARY:
A Drug-Drug Interaction study to assess the effects of itraconazole, carbamazepine and quinidine on the Pharmacokinetics and Safety of EDP-235.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP-235. A male participant who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection
* A positive urine drug screen at Screening or Day -1
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy)
* History of regular alcohol consumption
* Participation in a clinical trial within 30 days prior to the first dose of study drug
* For Part 2 participants:

  * Participants of Asian ancestry, given association of carbamazepine and severe rash (Stevens-Johnson Syndrome [SJS and Toxic Epidermal Necrolysis [TEN]) with HLA-B 1502 in this population
  * Platelets, white blood cell count or hemoglobin below the lower limit of normal, due to reported incidence of agranulocytosis and aplastic anemia with carbamazepine.
* For Part 2 and Part 3 participants, the following cardiovascular abnormalities:

  * QRS duration >110 ms
  * Incomplete right bundle branch block or any complete bundle branch block
  * Heart rate <40 or >90 beats per minute (per vital sign capture while rested)
  * History of unexplained syncope, structural heart disease, or clinically significant arrhythmias
  * Personal or family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome
  * PR interval >220 ms or any 2nd or 3rd degree AV block
  * Ventricular pre-excitation
* History of drug allergy to itraconazole or other azole antifungals; history of drug allergy to carbamazepine or carboxamide derivatives [e.g. oxcarbazepine]; known hypersensitivity to drugs structurally related to carbamazepine [e.g.: tricyclic antidepressants] or any of its excipients);history or known hypersensitivity to mefloquine, quinine, or quinidine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-235 with and without coadministration with Itraconazole | Day 1 through Day 19
AUC of EDP-235 with and without coadministration with Itraconazole | Day 1 through Day 19
Cmax of EDP-235 with and without coadministration with Carbamazepine | Day 1 through Day 26
AUC of EDP-235 with and without coadministration with Carbamazepine | Day 1 through Day 26
Cmax of EDP-235 with and without coadministration with Quinidine | Day 1 through Day 13
AUC of EDP-235 with and without coadministration with Quinidine | Day 1 through Day 13

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- ICON, plc., Lenexa, Kansas, United States